CLINICAL TRIAL: NCT01510730
Title: Effect of Helicobacter Pylori Eradication on the New Tumor Development After Endoscopic Resection of Gastric Tumors
Brief Title: Helicobacter Pylori Eradication After Endoscopic Resection of Gastric Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeongmin Choi, M.D., Seoul National University Hospital, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20052011
Record Dates: First submitted 2012-01-11; First posted 2012-01-16 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Gastric Tumor; Helicobacter Pylori; Endoscopic Resection; Metachronous Neoplasms
Keywords: gastric tumor; Helicobacter pylori; endoscopic resection; metachronous neoplasms
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms, Second Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): no treatment for Helicobacter pylori infection
- treatment group (Active Comparator): treatment group receive eradication treatment for helicobacter pylori infection
  Interventions: Drug: eradication treatment of Helicobacter pylori infection

INTERVENTIONS:
Drug: eradication treatment of Helicobacter pylori infection — Eradication group receive Omeprazole sodium 20mg, amoxicillin 1g, clarithromycin 500mg orally at the same time twice daily for 7 days.
  Arms: treatment group

SUMMARY:
The purpose of this study is to determine whether Helicobacter pylori eradication could reduce the new tumor development after endoscopic resection of gastric tumor.

DETAILED DESCRIPTION:
The association between Helicobacter pylori infection and development of gastric cancer has been established by epidemiologic studies. Conversely, eradication of H. pylori showed no significant reduction of the incidence of gastric cancer in a large-scale, double-blind, randomized controlled trial. Eradication of H. pylori to prevent cancer was only effective in the subgroup without precancerous lesions (i,e, dysplasia, intestinal metaplasia, and atrophy). In contrast, randomized prospective study in Japan showed that H. pylori eradication after endoscopic resection of early gastric cancer significantly reduced metachronous gastric cancer. To solve this conflicting issue is critical because gastric cancer is the second leading cancer incidence worldwide, particularly Korea, Japan, and China have highest cancer incidence, and its incidence might decrease by H. pylori eradication treatment.

With respect to therapeutic modality, endoscopic resection for early gastric cancer is currently the established treatment of choice in Korea and Japan because it has been proven to be both minimally invasive and effective in the curative treatment of early gastric cancer.

Endoscopic resection has also been performed in the gastric dysplasia because dysplasia has to some extent malignant potential although firm evidence is lacking. In comparison with surgical resection, endoscopic resection conserves remnant stomach. Accordingly, patients treated with endoscopic resection have higher possibility for metachronous gastric cancer than those treated with surgical resection.

So far, it has not yet been clearly established whether H pylori eradication for gastric tumors (early gastric cancer and gastric dysplasia) could reduce metachronous cancer. We performed randomized controlled, open-label trial on the effect of new cancer development after H pylori eradication for gastric tumors.

ELIGIBILITY:
Inclusion Criteria:

* H pylori infected patients with gastric low-grade dysplasia, high-grade dysplasia, and early gastric cancer
* Gastric tumor is completely removed through endoscopic resection.

Exclusion Criteria:

* Patients underwent gastrectomy before enrollment
* patients underwent endoscopic resection before enrollment
* Previous history of eradication for H. pylori
* Pregnancy
* Aged <20 yr old or aged >75 yr old
* Patients underwent additional gastrectomy due to incomplete endoscopic resection

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 855 (Actual)
Dates: Start 2005-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Effect of eradication of Helicobacter pylori on incidence of metachronous gastric carcinoma after endoscopic resection of gastric tumor. | we set the time frame as at least three years.
  Primary outcome is the incidence of new cancer development after endoscopic resection of gastric tumors between eradication and control groups. Previous reports showed the incidence of new cancer between two groups differs at least 3years.

SECONDARY OUTCOMES:
effect of eradication of Helicobacter pylori on incidence of High grade dysplasia development after endoscopic resection of gastric tumor. | 3 years
  Gastric high grade dysplasia has high malignant potential. Considering this, we set high grade dysplasia as secondary outcome measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Gyun Kim, professor, Principal Investigator — Department of Internal Medicine and Liver Research Institute
Locations (1):
- Department of Internal Medicine and Liver Research Institute, Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Choi JM, Kim SG, Choi J, Park JY, Oh S, Yang HJ, Lim JH, Im JP, Kim JS, Jung HC. Effects of Helicobacter pylori eradication for metachronous gastric cancer prevention: a randomized controlled trial. Gastrointest Endosc. 2018 Sep;88(3):475-485.e2. doi: 10.1016/j.gie.2018.05.009. Epub 2018 May 22. PMID 29800546
- [Derived] Choi J, Kim SG, Yoon H, Im JP, Kim JS, Kim WH, Jung HC. Eradication of Helicobacter pylori after endoscopic resection of gastric tumors does not reduce incidence of metachronous gastric carcinoma. Clin Gastroenterol Hepatol. 2014 May;12(5):793-800.e1. doi: 10.1016/j.cgh.2013.09.057. Epub 2013 Oct 5. PMID 24100112